CLINICAL TRIAL: NCT02591758
Title: Novel Vitality Indices Derived From the Hexoskin in Patients Affected With Angina Undergoing Coronary Revascularization or Medical Therapy (NOVA-SKIN Study)
Brief Title: Novel Vitality Indices Derived From the Hexoskin in Patients Affected With Angina Undergoing Coronary Revascularization or Medical Therapy
Acronym: NOVA-SKIN
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Marc Jolicoeur, Principal Investigator, Montreal Heart Institute
Other Study IDs: 2015-1919
Record Dates: First submitted 2015-10-09; First posted 2015-10-30 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Chronic Stable Angina
Keywords: Hexo-Skin; Hexoskin; NOVA-SKIN; angina; biometric vest
MeSH Terms: conditions — Angina, Stable; Angina Pectoris | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stable Angina with coronary angiogram: This study aims to correlate the biometric data collected and derived from the Hexoskin with the standard physiological assessment, in patients referred for coronary angiography for limiting angina. Afterwards, the clinician will decide of the best treatment strategy for the patient: coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) or no revascularization.
  Interventions: Device: Hexoskin Vest; Behavioral: Cardiac rehabilitation program; Other: Anxiety assessment as determined by the GAD-7; Other: Angina assessment with the angina diary, the SAQ and the SF-36; Other: Exercise stress test; Other: Holter monitoring

INTERVENTIONS:
Device: Hexoskin Vest — The Hexoskin vest will be used at home to monitor the patient before and after the coronary angiography, during a treadmill test and during a home cardiac rehabilitation program.
Behavioral: Cardiac rehabilitation program — A 6 sessions home cardiac rehabilitation program will be prescribed to the patient 2 to 4 weeks after the coronary angiogram. Those sessions will take place under Hexoskin surveillance. One session will take place at our specialized institution and six sessions will take place at home over the time span of two to three weeks.
Other: Anxiety assessment as determined by the GAD-7 — Anxiety assessment using the General Anxiety Disorder (GAD-7) scale, at the end of the study, to see if the Hexoskin relieved the anxiety patients can feel at home when exercising after a percutaneous coronary intervention.
Other: Angina assessment with the angina diary, the SAQ and the SF-36
  Other Names: Angina assessment with the angina diary, the Seattle Angina Questionnaire (SAQ) and the Short Form 36 (SF-36)
Other: Exercise stress test — Using the RAMP protocol before and after the coronary intervention, under Hexoskin surveillance.
Other: Holter monitoring — 24-hour Holter monitoring before and after the coronary angiogram with simultaneous Hexoskin reading.

SUMMARY:
The first and foremost manifestation of ischemic heart disease (IHD) is angina. At a global level, patients with chronic angina are at risk of poor vital status and deconditioning. Medical therapy and coronary revascularization using coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) can effectively relieve angina . In spite of all the available treatment options, the assessment of angina remains a challenge. Angina has a cyclical pattern and will naturally worsen and improve as days go by. Likewise, angina can be significantly biased by the placebo effect. Clinically angina is most frequently quantified with the Canadian Cardiovascular Society (CCS) classes system. In research protocols, angina is often quantified with health-related quality of life questionnaires and diaries. None of the tool available accounts for an important phenomenon called ischemic threshold adaptation, which could be defined as a limitation of their activity level under the ischemic level, which will translate into fewer angina episodes and a seemingly stable condition. Better clinical assessment tools that take into consideration the ischemic threshold adaption are needed.

Despite increased interest in wearable biometrics clothing in medicine, no prospective study has documented their utility to assess angina and to monitor the rehabilitation in cardiac patients. The Hexoskin™ is a biometric vest that can collect physiological data from individuals in their natural daily living environment. Currently, the use of biometric clothing is confined to a niche exploited exclusively by health enthusiasts, athletes or astronauts. As we enter this new age of virtual healthcare, tools like wearable biometrics could represent a giant leap forward in assisting healthcare professionals and patients. This will translate a better assessment of their health status, will allow physicians to target the right treatment strategy, ultimately improving case-selection and outcomes.

Our objective is to prospectively validate the wearable biometrics clothing Hexoskin™ against established standards used to assess chronic stable angina. In addition, the investigators want to derive a novel vitality index from the data generated by this device that will subsequently be used to propose a new angina classification system that will account for ischemic threshold adaptation. Moreover, the investigators want to evaluate the safety and efficacy of Hexoskin monitor patients undergoing home-based cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent form
2. Patient 18 years of age
3. History of coronary artery disease that consists of a well-documented medical history (over 3 months prior to the enrolment) of myocardial infarction or significant coronary artery disease with non-invasive angiographic confirmation.
4. Symptoms that support the diagnosis of chronic angina and/or a history of an abnormal exercise response limited by angina and/or electrocardiograph (ECG) changes.
5. All-comers with stable or unstable moderate-to-severe angina pectoris (Canadian Cardiovascular Class [CCS] II-III or IV subsequently medically stabilized (minimum 7 days) despite guideline directed medical therapy due to a reversible myocardial ischemia deemed sufficiently severe to justify a coronary angiography.
6. Patient can be treated percutaneously, surgically or medically.
7. Willing to undertake a cardiac rehabilitation program at home
8. Patient understands the nature of the device and is able to wear the Hexoskin for 24h Patient is willing to comply with specified follow-up evaluation and can be contacted by telephone.

Exclusion Criteria:

1. Recent (<1 week) acute coronary syndrome
2. Decompensated congestive heart failure (CHF) or hospitalization due to CHF during the 3 months prior to screening.
3. Severe valvular disease
4. High-risk criteria demonstrated on the treadmill stress test (Appendix D5)
5. With contraindications to, unable to, or with other co-morbidities that may prevent or interfere with the ability to perform treadmill stress test (including but not limited to : pulmonary hypertension, functionally limiting chronic obstructive pulmonary disease (COPD), history of pulmonary tuberculosis, prior hospitalization for acute exacerbation of chronic lung disease, home oxygen use, chronic oral steroid therapy that can limit exercise capacity, functionally limiting peripheral artery disease.
6. Patients for whom an home-based cardiac rehabilitation is contraindicated or not possible
7. Left ventricular ejection fraction (LVEF) < 40% or patients with defibrillator or cardiac resynchronisation pacemaker.
8. Severe left ventricular (LV) hypertrophy (defined as septal wall thickness at echocardiography of more than > 13 mm)
9. Congenital cardiac defects, severe uncontrolled hypertension (seated systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mm Hg), severe anemia, suspected or known dissecting aortic aneurysm, acute myocarditis or pericarditis, thrombophlebitis or pulmonary embolism.
10. Presence of electrocardiographic or other abnormalities/factors that could interfere with exercise electrocardiograph interpretation or may lead to a false positive stress test (See appendix B for more details)
11. Clinically significant arrhythmias, rapid atrial fibrillation (> 110 beats per minute at rest) or atrioventricular conduction block greater than first degree.
12. Planned need for concomitant cardiac surgery, such as valve surgery.
13. Refusal or an inability to perform cardiac rehabilitation.
14. Moribund patients, or patients with comorbidities limiting life expectancy < 1 year.
15. Any contra-indications to the treadmill stress test (See Appendix D6)
16. Mental condition (psychiatric or organ cerebral disease) rendering the subject unable to understand the nature, scope and possible consequences of the trial or mental retardation or language barrier such that the patient is unable to give informed consent.
17. Potential for non-compliance towards the requirements in the study protocol and/or follow-up visits
18. Any other conditions that, in the opinion of the investigator, are likely to prevent compliance with the study protocol or pose a safety concern if the subject participates in the study.
19. Currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty (30) subjects who meet all of the inclusion criteria and none of the exclusion criteria and who successfully wear the Hexoskin vest in the run-in will be eligible to study participation. Subjects will be recruited as outpatient, from the specialized angina clinic at the Montreal Heart Institute (MHI) or as an inpatient, after screening by the research team.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Validation of the Hexoskin measures : Average heart rate | Two months to three months
  Correlation between the heart rate as determined by the Hexoskin with the reference data provided by the Holter monitoring and treadmill stress test
Validation of the vitality index with angina class as assessed by the CCS Class | Two to three months
Validation of the vitality index with quality of life using the Seattle Angina Questionnaire | Two to three months
  The changes in the vitality index compared with changes quality-of-life as measured by the Seattle Angina Questionnaire
Validation of the vitality index with Anxiety using the GAD-7 | Two to three months
  The changes in the vitality index compared with changes of anxiety as measured by the General Anxiety Disorder Scale - 7 .
Validation of the vitality index with quality of life using the SF-36 | Two to three months
  The changes in the vitality index compared with changes quality-of-life as measured by the Short-Form 36 (SF-36).
Validation of the vitality index with Anxiety using the ASI-3 | Two to three months
  The changes in the vitality index compared with changes of anxiety as measured by the Anxiety Sensitivity Index (ASI-3)
Responsiveness to the revascularisation procedure or medical treatment | Two to three months
  Difference of the vitality index before and after the revascularisation procedure or medical treatment
Validation of the Hexoskin measures : Arrhythmia detection | Two to three months
  : Correlation between the arrhythmias as determined by the Hexoskin with the reference data provided by the Holter monitoring.
Adjusting of the different subdomains of SF-36, Seattle Angina Questionnaire, Treadmill length, CCS class and weekly angina count before and after the coronary angiogram for the vitality index | Two to three months
  Adjusting of the different subdomains of SF-36, Seattle Angina Questionnaire, Treadmill length, CCS class and weekly angina count before and after the coronary angiogram for the vitality index and comparison between the difference detected before & after compared to the unadjusted metrics

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | Two to three months
  Mortality, re-infarction, revascularization procedure, ventricular arrhythmias and re-hospitalisation for angina.
Safety outcomes of the Hexoskin (Allergies, Intolerance) | Two to three months
  Allergies, Intolerance
Resource utilisation : Any overnight hospital stay | Two to three months
  * Rehospitalisation: Any overnight stay at the hospital.
  * Coronary care unit admission: Any overnight stay at the coronary care unit.
  * Intensive care unit admission: Any overnight stay at the intensive care unit.
Medical contact (Number of phone calls or unplanned clinic or emergency visit to the physician per patient) | Two to three months
  Any phone call or unplanned clinic visit to a physician.
Remote signal transmission integrity | Two to three months
  o Defined as the number of seconds the Hexoskin does not transmit any interpretable data divided by the total time the Hexoskin has been worn.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Jolicoeur Jolicoeur, MD, M.Sc., MHS, Study Chair — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada